CLINICAL TRIAL: NCT06685640
Title: Evaluation of Clinical Success and Parental Satisfaction of Prefabricated Stainless Steel Crowns and Zirconia Crowns Applied to Primary Molar Teeth
Brief Title: Comparison of Clinical Success of Stainless Steel Crowns and Zirconia Crowns in Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Kadriye Görkem Ulu Güzel, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AADÜDHF 2023/36
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dental Caries; Pulpotomy
Keywords: primary molars; stainless steel crowns; zirconia
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prefabricated stainless steel crowns (Group A) (Experimental): Groups that received prefabricated stainless steel crowns
  Interventions: Other: prefabricated stainless steel crowns
- Prefabricated zirconia crowns (Group B) (Experimental): Groups that received prefabricated zirconia crowns
  Interventions: Other: prefabricated zirconia crowns

INTERVENTIONS:
Other: prefabricated stainless steel crowns — Full coverage restoration after pulpal treatment in multi-surface deep caries of primary mandibular second molars requiring pulpotomy
  Arms: prefabricated stainless steel crowns (Group A)
Other: prefabricated zirconia crowns — Full coverage restoration after pulpal treatment in multi-surface deep caries of primary mandibular second molars requiring pulpotomy
  Arms: Prefabricated zirconia crowns (Group B)

SUMMARY:
Evaluation and understanding of clinical success, parental satisfaction and effects on periodontal tissues are the main expected benefits of prefabricated zirconia crowns and prefabricated stainless steel crowns. For a long time, stainless steel crowns have been the restorative material of choice for children's primary and permanent posterior teeth. Today, prefabricated zirconia crowns are more popular than other options because they meet aesthetic expectations and have high mechanical strength. The aim of this study is to evaluate and compare the periodontal health, plaque accumulation, opposing tooth wear, parental satisfaction, and clinical performance (color match, retention, marginal integrity, marginal discoloration, anatomic form, secondary caries, surface roughness, surface gloss and postoperative sensitivity) of pediatric prefabricated stainless steel and zirconia crowns applied after pulpotomy to asymptomatic, multifaceted, deep carious primary mandibular second molars.

DETAILED DESCRIPTION:
MATERIALS AND METHODS/RESEARCH TECHNIQUES:

Material:

In the study, two different prefabricated crowns will be applied to the right and left primary mandibular second molars after pulpotomy using a split-mouth design. One will be a prefabricated zirconia crown and the other will be a prefabricated stainless steel crown. The sample size was calculated by G*Power analysis program as 12 teeth, 6 teeth in each group. Since this sample size would reduce the validity and reliability of future statistical tests, it was decided to conduct the study with a total of 20 samples, 10 in each group, taking into account possible data loss and the power of the study. Teeth will be randomly divided into two groups according to crown type.

The study will be terminated when the last visit of the last patient providing the sample is completed and the data is finalized.

Method:

* Before the treatment of primary mandibular second molars that meet the inclusion criteria, topical anesthesia (Vemcaine Pump Spray, VEM İlaç, Turkey) containing 10% lidocaine will be applied to the anesthesia area with a cotton pellet. After topical anesthesia, local anesthesia (Maxicaine Ampoule, VEM İlaç, Turkey) containing 40 mg articaine hydrochloride and 0.006 mg epinephrine hydrochloride in 1 ml will be administered.
* Then, the area will be cleaned under rubber dam isolation, and the coronal pulp will be removed. Hemostasis will be provided with a sterile cotton pellet moistened with serum for 5 minutes, and hemostasis will be achieved with ferric sulfate (ViscoStat™, Ultradent, Germany) for 15 seconds.
* The pulp chamber will be filled with MTA (NeoMTA Putty, NuSmile, TX, USA), then a 0.5 mm layer of resin-modified glass ionomer will be applied to the cavity floor, and the restoration will be completed with composite.
* The first step in applying stainless steel crowns will be to select the crown length. First, high-speed rotary tools will be used to prepare 1.5-2 mm occlusal reduction with diamond burs; a 1-2 mm subgingival preparation will be made from the gingival margin. The proximal surfaces will be reduced approximately 1 mm thick, starting from the occlusal and buccally, lingually, and gingivally from the mesial and distal contact points of the tooth.
* In order to achieve full adaptation to the tooth, after any necessary corrections, the crown edge will be curved with the help of forceps, and the edge will be trimmed with scissors or a bur until cervical adaptation is achieved. The shortened crown edges will be polished with the help of discs and rubbers.
* The teeth to be coated with zirconium will be prepared subgingivally from 2 mm occlusal and 1-2 mm from the gingival margin in accordance with the manufacturer's instructions.
* Since zirconia crowns are not flexible, the mesial and distal walls will be prepared parallel to the adjacent teeth, taking into account the distance to ensure passive adaptation.
* A conical diamond bur will be used in proximal reduction to ensure passive seating of the selected crown. The appropriate size crown will be found by trial.
* After the appropriate crown is selected for zirconia crowns, a cotton pellet moistened with sterile serum is applied to the area for 5 minutes to control bleeding, and the bleeding will be stopped. If necessary, bleeding control agents or retraction cords will be used to prevent active bleeding during cementation.
* The crowns in both groups are cemented with FujiCEM Evolve (GC, Tokyo, Japan). This cement in the RMCIS group is in paste form. It is applied directly into the crown in an injectable form with its own special tip and polymerized with a light device for 10 seconds. The cement residue accumulated at the gingival margin is cleaned with a probe, and a setting time of 4-5 minutes is waited in accordance with the manufacturer's instructions. Occlusion is checked. After the cementation is completed with the appropriate application technique, the cement residue accumulated at the gingival margin is cleaned with a probe tip. If a scratch occurs on the crowns during this process, this mark is cleaned with a bur, and the surface is polished with polishing discs.

In general, in the evaluation of success:

* Teeth that have been extracted due to abscess development in control appointments.
* Dissolution of cement and decementation of the crown.
* Internal and external root resorption seen in radiographic evaluation.
* Teeth with lesions in the furcation region.
* Teeth with widening in the periodontal ligament space will be evaluated as unsuccessful.

Plaque Index and Gingival Index in pediatric prefabricated stainless steel and zirconia crowns applied to asymptomatic primary mandibular second molars after pulpotomy will be evaluated at baseline and at the 1-month, 3-month, 6-month, and 12-month follow-ups. Tooth Wear Index, Modified United States Public Health Service (USPHS) Criteria, and parental satisfaction will also be assessed at the 1-month, 3-month, 6-month and 12-month follow-ups. Intraoral photographs will be taken immediately after treatment and at each follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* Age range of children from 4 to 5 years.
* Systemically healthy.
* Children who are positive and extremely positive according to the Frankl behavior scale.
* Asymptomatic primary mandibular second molars with multi-surface deep caries requiring pulpotomy treatment.
* No history of spontaneous pain.
* Primary mandibular second molars where bleeding at the pulpotomy site can be controlled within 3 to 5 minutes.
* Having opposing teeth in occlusal contact.
* Patients without any periodontal-related attachment loss.
* Patients without abscesses or fistulas on primary second molars.
* Children who verbally and in writing agree to participate in the study and are willing to attend regular follow-up appointments will be included.

Exclusion Criteria:

* Having a systemic disease.
* Periapical infection, abscess, or mobility in primary second molars.
* Those with active periodontal disease.
* Malocclusion or missing opposing tooth.
* Primary second molars with pathological internal or external resorption.
* Physiological root resorption exceeding 1/3 of the root.
* Children with bruxism or unilateral chewing habits will not be included in the study.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in periodontal health (Gingiva) | baseline, 1 months, 3 months, 6 months, 12 months
  Gingival evaluation of the patients will be made according to the Loe and Silness Gingival Index.
  According to this index system:
  0 : Normal (absence of inflammation)
  1. : Mild gingivitis (slight change in color, slight edema; no bleeding on probing)
  2. : Moderate gingivitis (redness, edema, and glazing; bleeding on probing)
  3. : Severe gingivitis (marked redness and edema; ulceration; tendency to spontaneous bleeding)
Change in periodontal health (Plaque) | baseline, 1 months, 3 months, 6 months, 12 months
  Plaque evaluation of the patients will be performed according to Silness and Loe Plaque Index. After the teeth isolated with cotton before the evaluation are air dried, the amount of plaque in the area near the gingival margin of each tooth will be examined by inspection and examination probe.
  According to this index system::
  0: No plaque.
  1. A thin layer of plaque is visible along the gingival margin. This thin layer can be detected with the examination probe.
  2. A moderate layer of plaque is visible along the gingival margin. This plaque can be visually detected.
  3. Heavy plaque accumulation is detected at the gingival margin and in the interdental area.
Wear of opposing natural teeth | 1 months, 3 months, 6 months, 12 months
  The Smith and Knight Tooth Wear Index classification, which is used to grade tooth wear, will be applied. The Smith and Knight Tooth Wear Index criteria are as follows: 0 Points (Buccal/lingual/occlusal/incisal): No loss of enamel surface characteristics (Cervical): No contour loss. Score 1 (Buccal/lingual/occlusal/incisal): Loss of enamel surface features (cervical): Minimal contour loss. Score 2 (Buccal/lingual/occlusal): Dentin opening with enamel loss of less than 1/3 of the surface (incisal): Dentin exposure with enamel loss (cervical): Less than 1 mm defect. Score 3 (Buccal/lingual/occlusal): More than 1/3 of the dentin surface exposed with enamel loss (incisal): Enamel loss and significant dentin loss (cervical): 1-2 mm defect. Score 4 (Buccal/lingual/occlusal): Complete loss of enamel or exposure of pulp/secondary dentin (incisal): Opening of pulp or secondary dentin (cervical): Defect larger than 2 mm or pulp/secondary dentin dehiscence.
Change in clinical performance | 1 months, 3 months, 6 months, 12 months
  Modified United States Public Health Service (USPHS) criteria will be used to evaluate color match, retention, marginal integrity, marginal discoloration, anatomic form, secondary caries, surface roughness, surface gloss and postoperative sensitivity. Restorations are evaluated and scored alphabetically. When evaluated in terms of any criterion; A: ideal restorations, B: restorations that are not ideal but within acceptable limits, C: restorations that are clinically unacceptable and need to be replaced, D: restorations that are already mobile or damage tissues receive a score of D. During clinical examination and recording, phonetically similar nomenclature is used to avoid misunderstanding of the score in terms of the letter pronounced by the physician: 'A'lfa, 'B'ravo, 'C'harlie, 'D'elta.

SECONDARY OUTCOMES:
Measuring of parental satisfaction | 1 months, 3 months, 6 months, 12 months
  Parental satisfaction will be evaluated on a five-point Likert scale, which responders specify their level of satisfaction.
  1. very dissatisfied
  2. dissatisfied
  3. neutrally satisfied
  4. satisfied
  5. very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Görkem Ulu Güzel, Doç. Prof., Study Director — Adnan Menderes Üniversitesi
Locations (1):
- Adnan Menderes University, Aydin, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data (IPD) will not be shared with other researchers